CLINICAL TRIAL: NCT04932239
Title: Effectiveness of Road Traffic Crashes First-aid Education on Knowledge, Attitude, and Practice Among Commercial Motorcyclists in Kigali-City, Rwanda
Brief Title: Effectiveness of Road Traffic Crashes First-aid Education Among Commercial Motorcyclists in Kigali-City, Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Christine UFASHINGABIRE MINANI, Principal investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JKEUPM-2021-173
Record Dates: First submitted 2021-05-28; First posted 2021-06-21 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: First Aid Education for Road Traffic Crashes
Keywords: Road traffic crashes; First aid education; knowledge,attitude and practice; motorcyclists
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: This study will be study will be a two-arms pre-post intervention study with a follow-up survey after 4 months
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Road traffic crashes first aid education module (Experimental): It is an education module aiming to address the topics related to first aid: Recognizing emergency, Call for help, Scene safety, Airway and breathing, Haemorrhage control, First aid kit, Immobilization of fractures and transport of injured people.
  Interventions: Other: first aid education
- Tuberculosis prevention education module (Placebo Comparator): This education module covers the definition of the disease, types ways of prevention in working place, and its management
  Interventions: Other: first aid education

INTERVENTIONS:
Other: first aid education — To teach commercial motorcyclists first aid for post-crash while waiting for medical team to reach the scene

SUMMARY:
Prehospital management after road traffic crashes(RTC) is a predicting factor to patient outcomes especially in Low-Income Countries where emergency medical services are lacking. This may explain the high mortality related to RTC in Rwanda for instance, where the delay to reach the hospital of these victims was found as an independent factor to death . For that reason, this study hypothesizes that the training of non -professionals as commercial motorcyclists could help to reduce trauma-related mortality and morbidity in Rwanda.

The protocol general objective is to evaluate the effectiveness of road traffic crashes first -aid education on knowledge, attitudes, and practice among commercial motorcyclists in Kigali-City, Rwanda.

Hypotheses are:

1. There is a difference in the baseline level of knowledge, attitudes, and practice on road crashes' first aid between the intervention and control groups of commercial motorcyclists.
2. There is a relationship between socio-demographic characteristics and knowledge, attitudes, and practice' levels on first aid among commercial motorcyclists.
3. There is a relationship between the education intervention and Knowledge, attitudes, and practice' level on first aid among commercial motorcyclists

DETAILED DESCRIPTION:
Specific objectives are:

1. To differentiate the baseline level of knowledge, attitudes, and practice on road crashes' first aid on the intervention and control groups of commercial motorcyclists.
2. To determine the relationship between socio-demographic characteristics of commercial motorcyclists and their level of knowledge, attitudes, and practice on first-aid.
3. To evaluate the effect of road traffic crashes' first-aid education on knowledge, attitudes, and practice of commercial motorcyclists after the intervention, within and between the intervention and control group.

   * Population: is the total number of commercial motorcyclists working in Kigali- City.
   * Sample size: The sample of 100 participants per group, i.e. intervention and control was estimated based on similar studies and using the following formula:

n = {[z(1-α/2) *√2 P̄ (1- P̄)] + [z(1-β)*√P1(1-P1) + P2 (1-P2)]}2 (P1-P2)2 The total number of participants is 200.

* Study instrument:self-administered questionnaire
* Intervention group will receive road traffic crashes' first aid education module
* Control group will get the Tuberculosis prevention in working place as an education module

Study procedure:

For the questionnaire, a pre-test on first aid will be done to the intervention and control groups before education intervention to measure the baseline level of knowledge attitudes and reported practice. In addition, a post-test immediately after education intervention will follow to assess the effectiveness of the educational intervention provided. The same evaluation will be conducted after four months of this training.

-Data analysis: SPSS version 25 will be used to analyze data. The first objective will be analyzed using descriptive statistics and chi-square. For the second objective, multiple logistic regression will be used to determine the relationship between socio-demographic characteristics and level of knowledge, attitude, and practice among commercial motorcyclists. Lastly, One way repeated ANOVA will be used to evaluate the relationship between first aid education intervention and level of knowledge, attitudes, and practice of commercial motorcyclists between pre and post-test scores. A P-value less than 0.05 will be considered statistically significant.

-Sensitivity analysis: Intention -to- treat( ITT) and per-protocol (PP) analyses will be used to determine the effect of dropout and non-response. The differences between the coefficients found from these two analyses will then calculated and stated as percentages.

* Ethical considerations:
* I got ethical approval from JKEUPM from Malaysia and IRB from Rwanda
* All study participants will provide informed consent prior to enrollment in the study. Data will be kept confidential and access will be restricted to the research team only. No participants' names will be required during data collection, only codes will be used.

Variables:

* Age
* Years of driving experience
* Level of education
* Previous training on first aid: will be measured by answering yes or no
* First aid education: refers to recognize the emergency, call for help, scene safety, airway, and breathing, hemorrhage control, first aid kit, immobilization of fractures, and transport of injured people.
* Knowledge: will be categorized into correct incorrect responses
* Attitudes: will be stratified into two groups: Strongly agree and agree will represent positive attitudes whereas unsure, disagree, and strongly disagree will stand for negative attitudes
* Practice: will refer to two clusters for correct and incorrect reported practices
* Intervention group: refers to a group of commercial motorcyclists that will receive road traffic crashes first aid education program
* Control group: is a group of commercial motorcyclists that will receive a placebo program concerning tuberculosis prevention in the working place

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a citizen of Rwanda and a commercial motorcyclist working in one of the Districts, Gasabo, Nyarugenge, and Kicukiro.
* Participant must have the age of 18 years and above.
* Participant must be able to read, write and speak Kinyarwanda (mother tongue)
* Participant must have at least a primary school level of education.
* Participant must have a motorcycle driving license.

Exclusion Criteria:

* Commercial motorcyclists with physical disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Change of knowledge on road traffic crashes first aid | immediate post intervention and after 4 months
  Knowledge outcome has ten close-ended questions assessing knowledge on first aid for road traffic crashes and each correct question will score one while the incorrect will score zero. Knowledge will be categorized into 3 categories:
  Good knowledge: refers to eight to ten correct answers out of ten. Fair knowledge: five to seven score out of ten whereas four and less out of ten is considered as low knowledge.
Change in attitudes on road traffic crashes first aid | immediate post interventions and after 4 months
  To assess attitudes, a five point likert scale on 7 questions will be done .( Strongly agree, agree , unsure, disagree ,and strongly disagree).
  Attitudes answers will be stratified into two groups: Strongly agree and agree will represent positive attitudes whereas disagree, unsure and strongly disagree will stand for negative attitudes
Change in reported practice toward first aid provision | immediate post interventions and after 4 months
  Regarding reported practice, four open questions will be given. The reported practice will refer to two clusters for correct and incorrect reported practices.

CONTACTS AND LOCATIONS:
Overall Officials: SOH KIM LAM, Prof., Study Chair — Universiti Putra Malaysia; KULANTHAYAN KC MANI, Prof., Study Director — Universiti Putra Malaysia; TWAGIRUMUGABE THEOGENE, Assoc. Prof., Study Director — Butare university Teaching Hospital; Rosliza Abdul Manaf, Assoc. Prof., Study Director — Universiti Putra Malaysia
Locations (1):
- University of Rwanda, Kigali, Kigali, Rwanda